CLINICAL TRIAL: NCT00782782
Title: Effect of Medications on Vascular Response in Patients With CHF and in Healthy Subjects
Brief Title: Vascular Sensitivity to Adrenergic Agonists in Patients With CHF and in Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Mordechai Muszkat, Hadassah University Hospital
Other Study IDs: 366-28.12.07
Record Dates: First submitted 2008-10-26; First posted 2008-10-31 (Estimated); Last update posted 2008-10-31 (Estimated); Status verified 2008-10

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples for norepinephrine and PRA will be retained
Oversight: Data Monitoring Committee: No

SUMMARY:
Congestive Heart failure (CHF) is asociated with changes in cardiac function and vascular responses. The aim of this study is to characterize these differences. Our hypothesis is, that there are differences in vascular responses between healthy subjects and patients with CHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congestive heart failure NYHA I-II
* Stable clinical condition

Exclusion Criteria:

* Resting systolic blood pressure < 100
* Resting heart rate < 50
* Hypersensitivity to dexmedetomidine, phenylephrine, isoproterenol, terbutaline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with congestive heart failure NYHA I-II and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
vascular sensitivity (ED50) and response (Emax) to dexmedetomidine, phenylephrine, isoproterenol and terbutaline | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Muszkat, Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel